CLINICAL TRIAL: NCT01233882
Title: An Open-Label, Single-Dose, Parallel-Group Study Of The Pharmacokinetics And Safety Of Bosutinib In Subjects With Renal Impairment And Matched Healthy Adults
Brief Title: Bosutinib In Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1871020
Record Dates: First submitted 2010-10-28; First posted 2010-11-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Renal Disease, End-Stage; Renal Insufficiency, Chronic; Renal Insufficiency, Acute
Keywords: Renal impairment; healthy volunteers
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Acute Kidney Injury; Renal Insufficiency | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy Volunteers (Experimental)
  Interventions: Drug: Bosutinib
- Mild Renal Impairment (Experimental)
  Interventions: Drug: Bosutinib
- Moderate Renal Impairment (Experimental)
  Interventions: Drug: Bosutinib
- Severe Renal Impairment (Experimental)
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — Single dose of 200 mg of bosutinib in subjects with normal renal function
  Arms: Healthy Volunteers
Drug: Bosutinib — Single dose of 200 mg of bosutinib in subjects with mild renal impairment
  Arms: Mild Renal Impairment
Drug: Bosutinib — Single dose of 200 mg of bosutinib in subjects with moderate renal impairment
  Arms: Moderate Renal Impairment
Drug: Bosutinib — Single dose of 200 mg of bosutinib in subjects with severe renal impairment
  Arms: Severe Renal Impairment

SUMMARY:
This is a two-staged study of a single dose of 200 mg of bosutinib given to subjects with renal impairment and matching healthy volunteers. In Stage 1, only subjects with severe renal impairment and subjects with normal renal function will be enrolled. Subjects with mild and moderate renal impairment will be enrolled in Stage 2 if the results from Stage 1 suggest a substantial difference in PK profiles between subjects with severe renal impairment and subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged 18 to 65.
* Adequate hepatic function.
* Documented creatinine clearance by Cockroft-Gault formula indicative of the respective level of renal impairment: Severe renal impairment (CrCl <30 mL/min/1.73m2), moderate renal impairment (30 ≤ CrCl ≤50 mL/min/1.73m2), mild renal impairment (50 < CrCl≤80 mL/min/1.73m2) and normal renal function (CrCl >80 mL/min/1.73m2).

Exclusion Criteria:

* Use of any investigational drug or biologic within 4 weeks prior to the screening visit of during the screening period.
* Ongoing treatment with Digoxin or strong CYP3A4 inhibitors or inducers.
* Uncontrolled hypertension (for renally impaired subjects only).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of bosutinib and its active metabolites will be measured, PK parameters (AUCinf, Cmax, AUClast, Tmax, t1/2, Cl/F and Vz/F) of bosutinib and its active metabolites will be calculated. | 11 days

SECONDARY OUTCOMES:
Safety endpoints to include adverse events, physical examination findings, changes in clinical laboratory test results including ECGs, and changes in vital signs | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Saint Paul, Minnesota

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1871020&StudyName=Bosutinib%20In%20Subjects%20With%20Renal%20Impairment